CLINICAL TRIAL: NCT00695643
Title: Double-blind, Randomized, Placebo-controlled, Parallel Group, Multi-centre Phase III Clinical Study on the Efficacy and Tolerability of Mesalazine Granules vs. Placebo for the Prevention of Recurrence of Diverticulitis
Brief Title: Mesalazine Granules vs. Placebo for the Prevention of Recurrence of Diverticulitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAG-37/DIV; 2007-000680-22 (EudraCT Number)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Mesalazine
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalazine — 3 g per day
  Arms: A
Drug: Placebo — 0 g per day
  Arms: B

SUMMARY:
The purpose of the study is to determine whether mesalazine granules compared to placebo is effective in prevention of recurrence of disease.

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate the superiority of mesalazine granules compared to placebo in terms of the primary efficacy variable proportion of recurrence-free patients within 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of left-sided uncomplicated diverticular disease confirmed by ultrasonography or computed tomography
* Presence of at least one diverticulum of the left colon
* Most recent attack of left-sided uncomplicated diverticulitis responding to antibiotics and/or dietary modification within the last 6 months
* C-reactive protein (CRP) > upper limit of normal (ULN) at the start of the most recent attack

Exclusion Criteria:

* Complicated diverticular disease
* Right-sided diverticulitis
* Previous colonic surgery
* Presence of symptomatic organic disease of the gastrointestinal tract
* Active colorectal cancer or a history of colorectal cancer
* Hemorrhagic diathesis
* Active peptic ulcer disease, local intestinal infection
* Asthma if careful medical monitoring is not ensured
* Abnormal hepatic function or liver cirrhosis
* Abnormal renal function

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Proportion of recurrence-free patients within 48 weeks | 48 weeks

SECONDARY OUTCOMES:
Time to recurrence
Occurrence of diverticulitis-associated fever | 48 weeks
Number of days with left lower quadrant pain | 48 weeks
Stool consistency | 48 weeks
Severity of diarrhea | 48 weeks
Quality of Life (QoL) | 48 weeks
Health assessment | 48 weeks
Assessment of efficacy by investigator and patient | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kruis, Professor, Principal Investigator — Evang. Krankenhaus Kalk, Medical department
Locations (1):
- Evang. Krankenhaus Kalk, Medical department, Cologne, Germany

REFERENCES:
- [Result] Kruis W, Kardalinos V, Eisenbach T, Lukas M, Vich T, Bunganic I, Pokrotnieks J, Derova J, Kondrackiene J, Safadi R, Tuculanu D, Tulassay Z, Banai J, Curtin A, Dorofeyev AE, Zakko SF, Ferreira N, Bjorck S, Diez Alonso MM, Makela J, Talley NJ, Dilger K, Greinwald R, Mohrbacher R, Spiller R. Randomised clinical trial: mesalazine versus placebo in the prevention of diverticulitis recurrence. Aliment Pharmacol Ther. 2017 Aug;46(3):282-291. doi: 10.1111/apt.14152. Epub 2017 May 23. PMID 28543263
- [Result] Gracie DJ, Ford AC. Editorial: mesalazine to prevent recurrent acute diverticulitis-the final nail in the coffin. Aliment Pharmacol Ther. 2017 Aug;46(4):461-462. doi: 10.1111/apt.14180. No abstract available. PMID 28707796
- [Result] Kruis W, Greinwald R. Editorial: mesalazine to prevent recurrent acute diverticulitis-the final nail in the coffin. Authors' reply. Aliment Pharmacol Ther. 2017 Aug;46(4):462-463. doi: 10.1111/apt.14193. No abstract available. PMID 28707787